CLINICAL TRIAL: NCT01544010
Title: Optimal TTM Tailoring for Population Cessation
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: DA023191-01A1
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Smoking Cessation
Keywords: Transtheoretical Model; Tailored Print Intervention; Population-based; Behavioral Intervention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- assessment only control group (No Intervention): Assessment at baseline, 12, and 24 months
- Minimal Stage Tailoring (Active Comparator): This group will receive a Stage-Tailored Manual at baseline. It will also get Stage Tailored Feedback Reports based on assessments at Baseline, 6, and 12 months. Outcomes will be assessed at 24 months.
  Interventions: Behavioral: Stage-Tailored Manual; Behavioral: Stage Tailored Feedback Report
- Moderate TTM Tailoring (Active Comparator): This group will receive a Stage-Tailored Manual at baseline. It will also get Moderate TTM-Tailored Feedback Reports, that is, integrated tailored feedback reports based on assessments of stage of change, decisional balance and temptations at Baseline, 6, and 12 months. Outcomes will be assessed at 24 months.
  Interventions: Behavioral: Stage-Tailored Manual; Behavioral: Stage Tailored Feedback Report; Behavioral: Moderate TTM-Tailored Feedback Report
- Full TTM tailoring (Active Comparator): This group will receive a Stage-Tailored Manual at baseline. It will also get Full TTM-Tailored Feedback Reports, that is, integrated tailored feedback reports based on assessments of stage of change, decisional balance (pros + cons), temptations and (ten) processes of change at Baseline, 6, and 12 months. Outcomes will be assessed at 24 months.
  Interventions: Behavioral: Stage-Tailored Manual; Behavioral: Stage Tailored Feedback Report; Behavioral: Moderate TTM-Tailored Feedback Report; Behavioral: Full TTM-Tailored Feedback Report
- Enhanced TTM+Addiction Tailoring (Active Comparator): This group will receive a Stage-Tailored Manual at baseline. It will also get Enhanced TTM+Addiction Tailored Feedback Reports, that is, integrated tailored feedback reports based on assessments of addiction levels (# cigarettes/day) stage of change, decisional balance (pros + cons), temptations and (ten) processes of change at Baseline, 6, and 12 months. Outcomes will be assessed at 24 months.
  Interventions: Behavioral: Stage-Tailored Manual; Behavioral: Stage Tailored Feedback Report; Behavioral: Moderate TTM-Tailored Feedback Report; Behavioral: Full TTM-Tailored Feedback Report; Behavioral: Enhanced TTM+Addiction Tailored Feedback Report

INTERVENTIONS:
Behavioral: Stage-Tailored Manual — Manual with 5 sections for each Stage of change delivered at baseline
  Other Names: Stage-based Manual; Stage-targeted self help manual
  Arms: Enhanced TTM+Addiction Tailoring; Full TTM tailoring; Minimal Stage Tailoring; Moderate TTM Tailoring
Behavioral: Stage Tailored Feedback Report — Tailored printed feedback reports based on assessments of stages of change were delivered at baseline, 6 months and 12 months.
  Other Names: Stage Targeted Feedback Report
  Arms: Enhanced TTM+Addiction Tailoring; Full TTM tailoring; Minimal Stage Tailoring; Moderate TTM Tailoring
Behavioral: Moderate TTM-Tailored Feedback Report — Tailored printed feedback report based on assessment of stages of change, Pros, Cons, and Temptations were delivered at baseline, 6 months and 12 months.
  Arms: Enhanced TTM+Addiction Tailoring; Full TTM tailoring; Moderate TTM Tailoring
Behavioral: Full TTM-Tailored Feedback Report — Tailored print feedback report based on assessment of Stages, Pros, Cons, Temptations, 10 Processes of Change were delivered at baseline, 6 months and 12 months.
  Arms: Enhanced TTM+Addiction Tailoring; Full TTM tailoring
Behavioral: Enhanced TTM+Addiction Tailored Feedback Report — Tailored print feedback report based on assessment of Addiction level (# cigarettes/day),Stages, Pros, Cons, Temptations, 10 Processes of Change were delivered at baseline, 6 months and 12 months.
  Arms: Enhanced TTM+Addiction Tailoring

SUMMARY:
This study explored optimal tailoring strategies for population tobacco cessation in 4 treatment groups and a control group over 24 months. Transtheoretical model (TTM) tailored feedback on all 14 variables has been found to be a robust population cessation strategy across studies. This proposal sought to find a subset of these variables that is optimal for tailoring, both minimizing response burden while maximizing effectiveness. Addiction variables have been demonstrated to predict smoking outcomes across studies as well, so we will integrate tailored feedback using TTM and addiction variables into an enhanced tailoring group. Optimally tailored feedback that both helps unmotivated smokers reduce their addiction and helps motivated smokers quit could lead to a breakthrough in population cessation.

DETAILED DESCRIPTION:
Smoking remains one of the biggest causes of premature morbidity and mortality. Nicotine addiction continues to challenge researchers to optimize their best interventions, and these challenges increase with efforts to integrate smoking cessation into multiple behavior change research and dissemination. Tailored intervention strategies have demonstrated effectiveness, yet much research remains to be done exploring optimal tailoring strategies. Transtheoretical model (TTM) tailored feedback on all 14 variables has been demonstrated to be a robust population cessation strategy across studies, producing 22-25% quit rates at 18-24 month final timepoints. This proposal sought to find a subset of these variables that is optimal for tailoring, both minimizing response burden while maximizing effectiveness. Addiction variables have been demonstrated to predict smoking outcomes across studies as well, so we will integrate tailored feedback using TTM and addiction variables into an enhanced tailoring group. Enhanced addiction tailored feedback that both helps unmotivated smokers reduce their addiction and helps motivated smokers quit could lead to a breakthrough in population cessation. This proposal tests four types of TTM-tailoring for smoking cessation in an additive design: assessment-only control group; Minimal tailoring (stage only); Moderate tailoring (stage, pros, cons, efficacy); Full TTM tailoring (all 14 TTM variables); and Enhanced TTM tailoring plus addiction variables. Smokers will be randomized to one of five treatment groups and evaluated at baseline, 6 months, 12 months, and 24 months. Treatment groups will receive tailored feedback at baseline, 6 months, and 12 months. Analyses will compare treatment groups on quit rates at the final timepoint to see how effectively each treatment helps smokers to quit. A series of mediation and moderation analyses will examine how each treatment works. This study has the potential to find an optimal tailoring strategy for population cessation that could accelerate future multiple behavior change research and dissemination efforts.

ELIGIBILITY:
Inclusion Criteria:

* smoker

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3006 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Smoking cessation (quit) rate | 24 months
  Self-report point prevalence abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A Redding, Ph.D., Principal Investigator — University of Rhode Island
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States

REFERENCES:
- [Background] Redding CA, Prochaska JO, Rossi JS, Kobayashi H, Yin HQ, Paiva AL, Velicer WF, Blaney C, Diamond E, Cottrill S. (2014). Levels of Transtheoretical Model Tailoring for Cessation: Randomized Trial Outcomes. Annals of Behavioral Medicine, 47, S238.